CLINICAL TRIAL: NCT02311335
Title: Genes Involved in Lipid Disorders
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150024; 15-H-0024
Record Dates: First submitted 2014-12-05; First posted 2014-12-08 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-06-23

CONDITIONS: Lipid Disorders
Keywords: Hypertriglyceridemia; Atherosclerosis; Genectic Variants; Hyperalphalipoproteinemia; Dyslipidemia; Natural History
MeSH Terms: conditions — Lipid Metabolism Disorders; Hypertriglyceridemia; Atherosclerosis; Cholesteryl Ester Transfer Protein Deficiency; Dyslipidemias

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Dyslipidemia patients

SUMMARY:
Background:

- Genes are the instructions our body uses to function. Researchers can look for changes, or variants, in the genes. The goal of this study is to find new gene changes that lead to lipid disorders. Older research methods looked at one or a few genes at a time. Genomic sequencing looks at most of the genes at once. Genomic sequencing may find the cause researchers haven t been able to find from past methods.

Objectives:

- To better understand genetic causes of lipid disorders through genomic sequencing.

Eligibility:

- People age 2 and older with unusual lipid disorders, and their relatives.

Design:

* Participants will be screened with a physical exam and medical history. They will have blood taken. They may give a saliva sample.
* Based on the screening test, researchers will chose 3-5 family members to perform the genomic sequencing. The sequencing will be done on a sample of DNA collected during the blood draw and saliva sample.
* Participants may be invited to take part in other protocols that may involve imaging of their heart or blood vessels. They do not have to participate. If they do, they will sign a separate consent for those tests.
* If a participant s family member cannot travel to the NIH, the NIH documents and consent will be reviewed during a teleconference. A blood or sputum kit will be mailed to them.

DETAILED DESCRIPTION:
The primary purpose of this discovery protocol is to identify new lipid genes from subjects with rare genetic lipids disorders. We will take advantage of the new technology of whole exome sequencing to find the cause of dyslipidemia that we haven t been able to find using past methods. We will work with geneticists to review the sequence data for unexpected gene changes (incidental findings) that do not explain the lipid disorder but gene changes that can cause medical disorders such as rare forms of cancer or heart disease. The opportunity to participate in the Clinical Center Genomics Opportunity (CCGO) program will enable us to take advantage of our expertise in other rare lipid disorders and translate this knowledge into new diagnostics and therapies, which is a key mission of the NIH.

ELIGIBILITY:
* INCLUSION CRITERIA:

Index cases to be included are those with unusual dyslipidemia. Relatives of affected individuals may also be included as appropriate.

Child Index: greater than or equal to 2 years older

Adult Index: greater than or equal to18 years older

Child relatives (siblings, cousins): greater than or equal to 2 years older

Adult Relative: greater than or equal to18 years older

(Biological parent, aunt, uncle or grandparent)

EXCLUSION CRITERIA:

1. Inability or unwillingness to provide informed consent or assent
2. Prisoners or other institutionalized persons will not be allowed to participate.
3. Children <2 years of age.

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Entire population.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2014-11-26 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Identify the gene(s) mutation (s) that causes rare cases of dyslipidemia | Ongoing
  Discovery data

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Shamburek, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The plan was not to share information because the groups were too small according to the rules and the information could lead to the identity of the subjects.

REFERENCES:
- [Background] Miller WG, Myers GL, Sakurabayashi I, Bachmann LM, Caudill SP, Dziekonski A, Edwards S, Kimberly MM, Korzun WJ, Leary ET, Nakajima K, Nakamura M, Nilsson G, Shamburek RD, Vetrovec GW, Warnick GR, Remaley AT. Seven direct methods for measuring HDL and LDL cholesterol compared with ultracentrifugation reference measurement procedures. Clin Chem. 2010 Jun;56(6):977-86. doi: 10.1373/clinchem.2009.142810. Epub 2010 Apr 8. PMID 20378768
- [Background] Oliveira MJ, van Deventer HE, Bachmann LM, Warnick GR, Nakajima K, Nakamura M, Sakurabayashi I, Kimberly MM, Shamburek RD, Korzun WJ, Myers GL, Miller WG, Remaley AT. Evaluation of four different equations for calculating LDL-C with eight different direct HDL-C assays. Clin Chim Acta. 2013 Aug 23;423:135-40. doi: 10.1016/j.cca.2013.04.009. Epub 2013 Apr 27. PMID 23628525
- [Background] Biesecker LG, Mullikin JC, Facio FM, Turner C, Cherukuri PF, Blakesley RW, Bouffard GG, Chines PS, Cruz P, Hansen NF, Teer JK, Maskeri B, Young AC; NISC Comparative Sequencing Program; Manolio TA, Wilson AF, Finkel T, Hwang P, Arai A, Remaley AT, Sachdev V, Shamburek R, Cannon RO, Green ED. The ClinSeq Project: piloting large-scale genome sequencing for research in genomic medicine. Genome Res. 2009 Sep;19(9):1665-74. doi: 10.1101/gr.092841.109. Epub 2009 Jul 14. PMID 19602640
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-H-0024.html